CLINICAL TRIAL: NCT02167789
Title: Clinical Evaluation of the Physiological Diagnosis Function in the PARADYM CRT
Brief Title: Clinical Evaluation of the Physiological Diagnosis Function in the PARADYM CRT Device
Acronym: CLEPSYDRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LivaNova (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ITSY02
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Heart Failure
Keywords: HF, diagnosis
MeSH Terms: conditions — Heart Failure; Disease

ARMS (1):
- PhD (No Intervention)
  Interventions: Device: Paradym CRT 8770

INTERVENTIONS:
Device: Paradym CRT 8770

SUMMARY:
This clinical investigation is a prospective, non-randomized, multi-center, pivotal trial.This trial is being performed in order to demonstrate the sensivity of the diagnostic feature "Physiological Diagnostic" (PhD).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the performance of a new sensor-based diagnostic feature, physiological Diagnostic (PhD)which as been implemented in the PARADYM CRT Cardiac Resynchronization System with defibrillation capabalities (PARADYM CRT System,model 8770.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible for implantation of a CRT-D device according to current available guidelines for cardiac resynchronization therapy
* Severe HF (NYHA Class III or IV) at the time of enrollment
* At least one HF-related event (as defined for primary objective) within the last 6 months before enrolment
* Subject continues to have heart failure symptoms despite receiving optimal medical therapy consistent with current practice guidelines for the pharmacological management of heart failure
* Scheduled for implant of a PARADYM 8770
* Signed and dated informed consent

Exclusion Criteria:

* Any contraindication for standard cardiac pacing
* Any contraindication for ICD therapy
* Abdominal implantation side
* Hypertrophic or obstructive cardiomyopathy
* Acute myocarditis
* Unstable coronary symptoms (unstable angina or myocardial infarction) within the last month
* Recent (within the last month) or planned cardiac revascularization or coronary angioplasty
* Correctable valvular disease that is the primary cause of heart failure
* Mechanical tricuspid valve
* Receiving continuous intra-venous infusion of positive inotropic therapy or intermittent therapy (intra-venous infusion) more than twice per week
* Heart transplant recipient
* Renal insufficiency requiring dialysis
* Already included in another clinical study
* Life expectancy less than 12 months
* Inability to understand the purpose of the study or refusal to cooperate
* Inability or refusal to provide informed consent and, if not part of the informed consent, a Health Insurance Portability and Accountability Act (HIPAA) authorization
* Unavailability for scheduled follow-up at the implanting center
* Known sensitivity to 1 mg dexamethasone sodium phosphate (DSP)
* Under guardianship
* Age of less than 18 years
* Pregnancy (Women of childbearing potential should have a negative pregnancy test prior to enrollment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2009-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Number of HF related events | 13 months

SECONDARY OUTCOMES:
Co morbidities | 13 months

CONTACTS AND LOCATIONS:
Locations (50):
- United States (5):
  - Dr. Haines, Kaplan, Phoenix,, Arizona
  - Drs. Lewis, Garg, Siegel, Phoenix,, Arizona
  - Drs. Jagmeet Singh, Kevin, Hiest, Boston, Massachusetts
  - Drs. John Fisher, Jay Gross, Montefiore, Bronx NY, New York
  - Dr. Gold, Charleston, South Carolina
- Canada (2):
  - Dr. Champagne, Dr. Philippon, Québec, Quebec
  - Drs. Thibualt, Guerra, Québec, Quebec
- France (15):
  - Dr. Dupuis, Angers, Angers
  - Dr. Defaye, Grenoble, Grenoble
  - Dr. Bru, La Rochelle, La Rochelle
  - Pr. Kacet, Lille, Lille
  - Dr. Pisapia, Marseille, Marseille
  - Pr. Davy, Montpellier, Montpellier
  - Dr. Burban, Nantes, Nantes
  - Dr Abbey, Nantes, Nantes
  - Dr. Ritter, Pessac, Pessac
  - Pr. Mabo, Rennes, Rennes
  - Pr. Anselme, Rouen, Rouen
  - Pr. Da Costa, Saint-Etienne, Saint Etienne
  - Dr. Delay, Toulouse, Toulouse
  - Pr. Sadoul, Vandœuvre-lès-Nancy, Vandoeuvre Les Nancy
  - Dr. Jauvert, Paris
- Germany (14):
  - Dr. Sperzel, Bad Nauheim, Bad Nauheim
  - Dr. Vogt, Bad Oeynhausen, Bad Oeynhausen
  - Dr. Butter, Bernau, Bernau
  - Pr. Brachmann, Coburg, Coburg
  - Dr. Klein - Dr. Oswald, Hanover, Hannover
  - Pr. Bauer, Heidelberg, Heidelberg
  - Pr. Mewis - Pr. Fröhlig, Homburg, Homburg
  - Dr. Wieckhorst, Kiel, Kiel
  - Dr. Bonnemeier, Lübeck, Lübeck
  - Pr. Weiss, Lüneburg, Lüneburg
  - Dr. Kolb, München, Munchen
  - Pr. Eckhardt, Münster, Münster
  - Dr. Fleck - Dr. Goetze, Berlin, State of Berlin
  - Dr. Schlegl, Berlin, State of Berlin
- Italy (2):
  - Dr. Leonardo Calo, Roma, Roma
  - Dr Mantovan, Treviso, Treviso
- Dr. Delnoy, Zwolle, Zwolle, Netherlands
- Spain (4):
  - Dr. Martinez, Alicante, Alicante
  - Dr. Brugada, Barcelona, Barcelona
  - Dr. Peinado, Madrid, Madrid
  - Dr. Beiras, Vigo, Vigo
- Dr Auricchio, Lugano, Lugano, Switzerland
- United Kingdom (6):
  - Dr. Leyva, Birmingham, Birmingham
  - Dr Fluck - Dr. Beeton, Chertsey, Chertsey
  - Dr. NG, Leicester, Leicester
  - Dr. Murgatroyd, London, London
  - Dr. Bowes, Sheffield, Sheffield
  - Dr. Morgan, Southampton, Southampton